CLINICAL TRIAL: NCT06789354
Title: Body Awareness and Perception Across Menstrual Phases: A Multidimensional Perspective
Brief Title: Body Awareness and Perception Across Menstrual Phases:
Status: Completed | Type: Observational
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Other Study IDs: 27.02.2020/29
Record Dates: First submitted 2025-01-13; First posted 2025-01-23 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2024-12

CONDITIONS: Menstrual Cycle
Keywords: Body Awareness; Menstrual Cycle
MeSH Terms: interventions — Surveys and Questionnaires; Restraint, Physical

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Female volunteers aged 18-35 years with regular menstrual cycles
  Interventions: Other: Questionnaire and Physical Exam

INTERVENTIONS:
Other: Questionnaire and Physical Exam — All assessments were carried out face-to-face with the same physiotherapist.

SUMMARY:
The study explores the dynamic interplay between body awareness and body perception across the menstrual cycle's phases, emphasizing hormonal influences on these dimensions. Conducted with 43 female participants aged 18-35, this research highlights significant variability in body-related experiences tied to hormonal fluctuations.

The study aims to address the gap in understanding how menstrual cycle phases impact women's body awareness-sensitivity to physiological states-and body perception, encompassing self-image and physical self-evaluation.

DETAILED DESCRIPTION:
Methods: Participants were divided based on menstrual phases: follicular, ovulatory, and luteal. Hormonal fluctuations were tracked through menstrual calendars and ovulation kits. Tools such as the Body Awareness Questionnaire (BAQ) and Multidimensional Body-Self Relations Questionnaire (MBSRQ) assessed participants' awareness and perception. Other assessments included the Premenstrual Syndrome Scale (PMS), Menstruation Attitude Scale (MAS), and physical activity tracking through the IPAQ-SF questionnaire.

Limitations The reliance on self-reported data and single-cycle assessments are noted as constraints, suggesting the need for longitudinal studies for greater robustness.

ELIGIBILITY:
Inclusion Criteria:

* female volunteers
* aged 18-35 years
* regular menstrual cycles

Exclusion Criteria:

* not using hormonal contraceptives in the preceding six months
* having no history of gynecological disorders
* having no chronic diseases

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — the research based on menstrual cycle.
Study Population: Female volunteers aged 18-35 years with regular menstrual cycles (28 ± 2 days) participated in the study,
Sampling Method: Probability Sample
Enrollment: 147 (Actual)
Dates: Start 2020-05-23 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2024-12-29 (Actual)

PRIMARY OUTCOMES:
Body Awareness Questionnaire (BAQ) | through study completion, an average of 1 year
  The Body Awareness Questionnaire (BAQ) is a self-assessment tool consisting of 18 items divided into four subscales (16). These subscales evaluate attentiveness to (1) bodily processes, including changes and reactions in the body, (2) the sleep-wake cycle, (3) the ability to predict the onset of illness, and (4) the prediction of bodily reactions. The questionnaire employs a 7-point Likert scale for scoring, where higher scores reflect greater body awareness. The BAQ has a total possible score ranging from a minimum of 18 to a maximum of 126. The Turkish adaptation of the BAQ, including validity and reliability analyses, was conducted by Karaca and Bayar, ensuring its applicability in Turkish-speaking populations (17).
Body Perception Scale (BPS) | through study completion, an average of 1 year
  The Multidimensional Body-Self Relations Questionnaire (MBSRQ), developed by Cash, is a self-report Likert-type scale designed to assess the structure of body image and attitudinal components of self-perception (18). The original instrument comprises 69 items, which evaluate three psychological dimensions characterized by emotional, cognitive, and behavioral traits, as well as three physical dimensions: physical appearance, physical competence, and biological integrity. The cognitive and behavioral aspects were subsequently consolidated under the category of 'orientation,' resulting in six distinct subscales within the questionnaire. An additional subscale, 'satisfaction with body domains,' was later introduced, bringing the total to seven subgroups. Lower mean scores on the MBSRQ indicate the presence of body image disturbances, providing valuable insights into individuals' attitudes and perceptions toward their bodies (18,19

CONTACTS AND LOCATIONS:
Locations (1):
- Marmara University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
I do not prefer